CLINICAL TRIAL: NCT01425242
Title: An Open-label PET-observer-blinded Pilot Study of the Effect of Aliskiren- Versus Amlodipine-based Antihypertensive Treatment in Patients With Small Abdominal Aortic Aneurysm and Mild to Moderate Hypertension on Aneurysmal FDG-uptake
Brief Title: Study on Anti-inflammatory Effect of Anti-hypertensive Treatment in Patients With Small AAA's and Mild Hypertension
Acronym: PISA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of participants
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jan D. Blankensteijn, Prof. Dr., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAA-PET/CT vumc; 2011-000538-12 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension; Abdominal Aortic Aneurysm
Keywords: inflammation; aneurysm; hypertension; aliskiren
MeSH Terms: conditions — Hypertension; Aortic Aneurysm, Abdominal; Inflammation; Aneurysm | interventions — aliskiren; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren (Experimental): Half of all subjects with mild to moderate hypertension and a small abdominal aortic aneurysm are treated with aliskiren, combined with hydrochlorothiazide if hypertension cannot be treated sufficiently with aliskiren monotherapy
  Interventions: Drug: Aliskiren
- Amlodipine (Active Comparator): Half of all subjects with mild to moderate hypertension and a small abdominal aortic aneurysm are treated with amlodipine, combined with hydrochlorothiazide if hypertension cannot be treated sufficiently with amlodipine monotherapy
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Aliskiren — Starting dose: Aliskiren 150 mg p.o, if hypertension is insufficiently treated Hydrochlorothiazide 12.5 mg p.o. tablet once daily for maximally 12 months can be added, the next step is to add increase the dosage of Aliskiren to 300 mg p.o. tablet once daily until maximally 12 months after baseline, the final step to take in case hypertension is still present is to increase Hydrochlorothiazide to 25 mg p.o. tablet once daily until maximally 12 months after baseline.
  Other Names: Rasilez
  Arms: Aliskiren
Drug: Amlodipine — Starting dose: amlodipine 5 mg p.o, if hypertension is insufficiently treated Hydrochlorothiazide 12.5 mg p.o. tablet once daily for maximally 12 months can be added, the next step is to add increase the dosage of amlodipine to 10 mg p.o. tablet once daily until maximally 12 months after baseline, the final step to take in case hypertension is still present is to increase Hydrochlorothiazide to 25 mg p.o. tablet once daily until maximally 12 months after baseline.
  Other Names: Norvasc
  Arms: Amlodipine

SUMMARY:
Inflammation of the blood vessel plays an important role in the development and growth of a dilated abdominal aorta. An elevated blood pressure leads to an increase in inflammation, therefore blood pressure lowering is an important part of the treatment of patients with a dilated abdominal aorta who also have an elevated blood pressure. In the investigators study the investigators compare the anti-inflammatory effects of 2 different blood pressure lowering strategies. The investigators hypothesize that both strategies will decrease inflammation, however the investigators believe the total decrease of inflammation depends on the type of blood pressure lowering medication used.

DETAILED DESCRIPTION:
Standard therapy of small AAAs currently consists of "watchful waiting" strategy with aggressive blood pressure control "Watchful waiting" includes an Ultrasound (more recently CT or MRI scan) every 12 months (for AAAs between 3.5 - 4.4 cm) or every 6 months (for AAAs between 4.5 and 5.5 cm) to observe. A growth rate of >7 mm/ 6 months has been suggested as a threshold for proceeding to aneurysm repair irrespective of aneurysm size. Clearly, there is need for a more sensitive method to evaluate the progress of AAA growth.

Recent publications have shown that evaluation of AAAs using FDG-uptake with PET-scan may identify small AAAs that are more prone to grow and/or rupture, as these AAAs as compared to normal aorta's show increased inflammatory activity , which is considered the major pathophysiological pathway. Evaluation of FDG-uptake is also sensitive enough to observe the short-term effects of endovascular intervention of large AAAs, as unpublished data show a statistically significant reduction in aneurismal FDG-uptake only 6 weeks after endovascular repair of large AAAs. Therefore, the change in aneurismal FDG-uptake may also be a very promising and sensitive method to evaluate treatment effects of medical interventions within a relatively short period of time (3 months).

Just as pressure unloading may represent an anti-inflammatory mechanism in endovascular repair of more advanced aneurysms, so may milder pressure unloading in moderately hypertensive individuals with smaller aneurysms display similar anti-inflammatory effects. Such a mild form of pressure unloading may be attainable with adequate anti-hypertensive drug therapy. In this context, however, a possible additional benefit may be that some anti-hypertensive drug classes have been proposed to exert specific anti-inflammatory effects relevant to aneurysm inflammation.

Local activation of multiple components of the renin angiotensin system has been implicated in both the development of aneurysms, as well as in their inflammatory component. In accordance, preliminary evidence from murine studies suggest that ACE inhibitors, for example, may reduce inflammatory activity in aneurysmatic vessel walls. However, since ACE inhibitors block the renin angiotensin system halfway it's path, and non-ACE conversion of angiotensin I occurs, a rationale exists to block the renin angiotensin system upstream of ACE. Upstream blockade of the renin-angiotensin system may have additional advantages in antagonising direct pro-inflammatory effects of renin itself, which have been identified in, for example, kidney tissue and retinal microvessels.

A case can thus be made for renin inhibition as a potential optimal strategy for reducing aneurysm inflammation in hypertensive patients with aortic aneurysms. In the proposed pilot trial, the direct renin inhibitor Aliskiren will be evaluated. As a control condition, an antihypertensive agent without postulated specific anti-inflammatory effects is appropriate. Calcium channel blockers represent such a class.

The current study will explore what the size and variability of the effect of aliskiren monotherapy, the combination of aliskiren/hydrochlorothiazide, amlodipine monotherapy, or the combination of amlodipine/hydrochlorothiazide on FDG-uptake is (if at all measurable on top of the effect of antihypertensive and statin therapy). This will allow more accurate power calculation of larger future studies aiming at prevention of AAA-progression (diameter and rupture).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a proven AAA of >30 mm and < 55 mm
2. Age between 18 and 75y (both inclusive)
3. Weight > 50 kg
4. Mild to moderate hypertension (defined as 130 < msSBP < 180 or 85< msDBP <110), at screening and/or baseline, without current antihypertensive medication.

Exclusion Criteria:

1. Patients without an AAA, or with an AAA ≥ 55 mm, or ≤ 30 mm
2. Patients with an AAA who are eligible for surgical repair for any reason
3. Diabetes mellitus
4. Inability of the subjects to switch from all prior antihypertensive medications safely as required by the protocol and need for drugs other than study drugs at the time of baseline
5. Severe hypertension (msSBP ≥180 mmHg and/or msDBP ≥110 mmHg) at screening and/or baseline
6. Pregnant or nursing (lactating) women
7. Known or suspected contraindications, including history of allergy or hypersensitivity (such as angioedema) to DRIs, CCBs, ACEIs, statins, acetylsalicylic acid or diuretics in general (for example, to aliskiren / amlodipine / hydrochlorothiazide / statins)
8. Concomitant drugs that are strong inhibitors of CYP3A4 or P-glycoprotein inhibitors (ketoconazole, itraconazole, nefazodone, clarithromycin, ritonavir, nelfinavir, cyclosporine, verapamil, quinidine)
9. Previous or current diagnosis of heart failure (NYHA Class II-IV)
10. Second or third degree heart block without a pacemaker, or potentially life-threatening arrhythmia during the 12 months prior to screening
11. Clinically symptomatic valvular heart disease at screening visit
12. A past medical history of clinically significant ECG abnormalities
13. Confirmed serum potassium ≥5.3 mEq/L (mmol/L) at screening or baseline.
14. Impaired renal function, defined as eGFR < 45 mL/min/1.73 m2 MDRD
15. Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation
16. Participation in any clinical investigation within four (4) weeks prior to first dose or longer if required by local regulations, and for any other limitation of participation based on local regulations.
17. Patients who have undergone prior radionuclide treatment or examinations or X-ray examinations with a cumulative radiation exposure, which added to the radiation exposure of the current study, would exceed local limits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in aneurysmal vessel wall inflammation | 3 months and 12 months
  Change from baseline in aneurismal FDG-uptake as measured with PET-CT after 3 and 12 months

SECONDARY OUTCOMES:
Change in abdominal aortic aneurysm diameter | 12 months
  Change from baseline in aneurismal diameter after 12 months
Change in large vessel inflammation | 3 months and 12 months
  Change from baseline in FDG-uptake in other large blood vessels after 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan D Blankensteijn, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands